CLINICAL TRIAL: NCT06814067
Title: Phase II Multicentered Study of Perioperative Ivonescimab Versus Pembrolizumab Combined with Standard of Care (SOC) in Patients with Resectable, Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Phase II Multi-centered Study of Perioperative Ivonescimab Versus Pembrolizumab Combined with Standard of Care (SOC) in Patients with Resectable, Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yu Wang, M.D., Professor, Chief of the department of head and neck surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Insight-4
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma HNSCC
Keywords: Neoadjuvant therapy; Immunotherapy; Ivonescimab; pembrolizumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Surgical Procedures, Operative; Radiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perioperative pembrolizumab (Active Comparator): Neoadjuvant pembrolizumab two cycles, followed by radical surgery. Adjuvant radiation/chemoradiation was decided based on pathologic risk factors. Then maintenance therapy of pembrolizumab for fifteen cycles was given.
  Interventions: Drug: Pembrolizumab; Procedure: Surgery; Radiation: Adjuvant radiotherapy
- Perioperative Ivonescimab (Experimental): Neoadjuvant ivonescimab two cycles, followed by radical surgery. Adjuvant radiation/chemoradiation was decided based on pathologic risk factors. Then maintenance therapy of ivonescimab for fifteen cycles was given.
  Interventions: Drug: Ivonescimab; Procedure: Surgery; Radiation: Adjuvant radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab — Two cycles of neoadjuvant pembrolizumab (200mg q3w) followed by radical surgery. Adjuvant radiotherapy/chemoradiotherapy is decided based on pathological risk factors. Fifteen cycles of pembrolizumab (200mg q3w)maintenance therapy was given.
  Arms: Perioperative pembrolizumab
Drug: Ivonescimab — Two cycles of neoadjuvant Ivonescimab (10mg/kg q3w) followed by radical surgery. Adjuvant radiotherapy/chemoradiotherapy is decided based on pathological risk factors. Fifteen cycles of Ivonescimab maintenance therapy (10mg/kg q3w) was given.
  Arms: Perioperative Ivonescimab
Procedure: Surgery — Radical surgery
Radiation: Adjuvant radiotherapy — Adjuvant radiotherapy with/without concurrent cisplatin-based chemotherapy, based on pathologic risk factors.

SUMMARY:
Head and neck squamous cell carcinoma (HNSCC) is one of the common malignant tumors in the world. More than 60% of HNSCC patients are locally advanced when first diagnosed. The treatment effect of locally advanced HNSCC is not ideal. About 50-60% of patients will have local recurrence within 2 years, and 20-30% of patients will have distant metastasis. The 5-year disease control rate is approximately 40%, and the 5-year overall survival rate is less than 50%.

In recent years, PD-1 inhibitors have shown significant efficacy in recurrent/metastatic HNSCC. The Keynote 040 and Checkmate 141 studies established the status of PD-1 inhibitors as second-line treatment in recurrent/metastatic HNSCC. The Keynote 048 study further established the value of PD-1 inhibitors alone or in combination with chemotherapy in the first-line treatment of recurrent/metastatic HNSCC. An increasing number of studies have attempted to explore the value of neoadjuvant therapy with PD-1 inhibitors in locally advanced HNSCC. For example,The Checkmate 358 study showed that the clinical objective response rate of neoadjuvant nivolumab monotherapy was 10.2%, and the major pathological response rate (MPR) was 2.9%.

Ivonescimab is a new PD-1/VEGF bispecific antibody drug, which can block both the PD-1 pathway and the VEGF pathway. This dual blocking mechanism is expected to enhance the efficacy of immunotherapy by improving the tumor microenvironment. Ivonescimab has been studied in Phase II to Phase III clinical studies in multiple tumor types such as lung cancer, breast cancer, and head and neck squamous cell carcinoma. For example, the HARMONi-2 study showed that ivocilizumab monotherapy had significantly better progression-free survival (PFS) than pembrolizumab in the treatment of PD-L1-positive locally advanced or metastatic non-small cell lung cancer (NSCLC). In recurrent and metastatic HNSCC, Ivonescimab alone or in combination with the CD47 monoclonal antibody Ligufalimab has better objective response rate (ORR) and disease control rate (DCR) than pembrolizumab.

The aim of this study is to compare the efficacy and safety of perioperative treatment with Ivonescimab and pembrolizumab in surgically resectable locally advanced head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. ) Patients who signed the informed consent and were willing to complete the study according to the protocol.
2. ) Age ≥18.
3. ) Patients diagnosed with head and neck squamous cell carcinoma by histology, including those with primary lesions in the oropharynx, oral cavity, larynx, or hypopharynx, or those with head and neck squamous cell carcinoma of unknown primary lesion after comprehensive examination and multidisciplinary discussion.
4. ) Locally advanced head and neck squamous cell carcinoma that can be surgically resected ( AJCC staging 8th edition: stage III-IVB), excluding T4b.
5. ) There was at least one measurable lesion before treatment, which met the requirement of " measurable lesion " in RECIST 1.1 standard.
6. ) Expected survival period: >3 months.
7. ) ECOG score 0-1.
8. ) Good organ function: Meet the following requirements:

   1. Absolute neutrophil count ( ANC ) ≥ 1.5 ×10 9 / L ;
   2. Platelet count ≥ 100 × 10 9 / L ;
   3. Hemoglobin ≥ 9 g/ dL ;
   4. Serum albumin ≥ 2.8 g/ dL ;
   5. Total bilirubin ≤ 1.5 × ULN , ALT , AST and / or ALP ≤ 2.5 × ULN ;
   6. Serum creatinine ≤ 1.5 × ULN and creatinine clearance ≥60 mL/min (Cockcroft-Gault );
   7. Activated partial thromboplastin time ( APTT ) and international normalized ratio ( INR ) ≤ 1.5 × ULN (screening is allowed for patients who are using stable doses of anticoagulant therapy such as low molecular weight heparin or warfarin and whose INR is within the expected therapeutic range of the anticoagulant ).
9. ) Patients with hepatitis B virus ( HBV ) infection and inactive / asymptomatic HBV carriers, or patients with chronic or active HBV , will be allowed to enroll if HBV DNA <500 IU/mL (or 2500 copies/mL ) at screening . Patients with positive hepatitis C antibodies will be allowed to enroll if HCV-RNA is negative at screening .
10. ) Women of childbearing age , who must have a negative urine or serum pregnancy test result within 7 days before treatment . They must use a medically approved contraceptive method (such as intrauterine device, contraceptive pills or condoms) during the study treatment, at least 3 months after the last use of immunotherapy and at least 6 months after the last use of chemotherapy.
11. ) Male subjects who are not sterilized must be willing to use a medically approved contraceptive method (such as intrauterine device, birth control pills or condoms) during the study treatment, at least 3 months after the last use of immunotherapy, and at least 6 months after the last use of chemotherapy.

Exclusion Criteria:

1. Patients who have had or are suffering from other malignant tumors in the past (except for those who have been cured and have survived cancer-free for more than 5 years, such as basal cell carcinoma of the skin, carcinoma in situ of the cervix, and papillary thyroid carcinoma).
2. Received any of the following treatments:a. Received any investigational drug within 4 weeks before the first use of the investigational drug; b. Enrolled in another clinical study at the same time, unless it is an observational (non-interventional) clinical study; c. Subjects who need to be given corticosteroids (≥ 10 mg prednisone equivalent per day) or other immunosuppressants for systemic treatment within 2 weeks before the first use of the study drug, except for the use of corticosteroids for local inflammation and prevention of allergies, nausea and vomiting. Other special cases need to be communicated with the investigator. In the absence of active autoimmune diseases, inhaled or topical steroids and adrenal cortical hormone replacement with a dose of ≥ 10 mg/ day prednisone efficacy dose are allowed; d. Those who have received anti-tumor vaccines or have received live vaccines within 4 weeks before the first administration of the study drug (if the new coronavirus vaccine is received, the interval between the vaccination and treatment must be more than 2 weeks) .
3. Uncontrolled cardiac clinical symptoms or diseases, such as: a. NYHA grade II or above heart failure; b. Unstable angina; c. Myocardial infarction within 1 year; d. Patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention.
4. Severe infection ( CTCAE > 2 ) occurred within 4 weeks before the first use of the study drug , such as severe pneumonia, bacteremia, infectious complications requiring hospitalization, etc.; baseline chest imaging examination indicated active lung inflammation, symptoms and signs of infection within 4 weeks of the first use of the study drug, or the need for oral or intravenous antibiotic treatment.
5. Patients with active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); but excluding autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone; type 1 diabetes using stable doses of insulin; patients with vitiligo or healed childhood asthma / allergy who do not require any intervention as adults.
6. Have a history of immunodeficiency, including positive HIV test, or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation and allogeneic bone marrow transplantation.
7. A history of interstitial lung disease (excluding radiation pneumonitis without hormone treatment) or non-infectious pneumonia.
8. Patients with active pulmonary tuberculosis infection found through medical history or CT examination, or patients with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or patients with a history of active pulmonary tuberculosis infection more than 1 year ago but without formal treatment.
9. Subjects have active hepatitis B ( HBV DNA ≥ 500 IU/mL or 2500 copies/mL ), hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the detection limit of the analytical method).
10. Underwent major surgery or severe trauma in the past 30 days.
11. The researcher assesses that the patient has a high risk of bleeding (such as a history of severe bleeding tendency or abnormal coagulation function, such as the tumor enveloping the carotid artery >180 degrees, the tumor invading the trachea, etc.).
12. Known history of psychotropic substance abuse, alcoholism or drug abuse.
13. Pregnant or breastfeeding women.
14. The researcher judges that the subject has other factors that may force him/her to terminate the study midway, such as other serious diseases (including mental illness) requiring combined treatment, serious abnormal laboratory test values, family or social factors that may affect the safety of the subject or the collection of trial data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2029-02-10 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Major pathological response | 4 months
  Major pathologic response, defined as ≤10% residual viable tumor in the resected primary tumor and lymph node tissue

SECONDARY OUTCOMES:
Event-free survival rate | One year
  Event free survival, defined as the time from the randomization to the first occurrence of any of the following events-disease progression that precludes surgical treatment, local recurrence or distant metastasis, or death from any cause. The Kaplan Meier method was used to estimate the EFS rate for each treatment group at 1 year after treatment assignment.
Overall survival rate | One year
  Overall survival, defined as the time from randomization to death from any cause. The Kaplan Meier method was used to estimate the OS rate for each treatment group at 1 year after treatment assignment.
pCR rate | 4 months
  Pathologic complete response rate, defined as no residual tumor within the resected primary disease and lymph node tissue.
Overall response of neoadjuvant therapy | 8 weeks
  Neoadjuvant treatment objective response rate (ORR), defined as the proportion of CR and PR subjects in each treatment group who took at least one cycle of neoadjuvant treatment, per RECIST 1.1 criteria.
Adverse event | From the time of randomization to 90 days after the last dose of immunotherapy.
  AE refers to an adverse medical event that occurs after a clinical trial subject receives a drug, but it is not necessarily causally related to the treatment. AE can be any unfavorable and unexpected symptoms, signs, laboratory abnormalities or diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wise-Draper TM, Gulati S, Palackdharry S, Hinrichs BH, Worden FP, Old MO, Dunlap NE, Kaczmar JM, Patil Y, Riaz MK, Tang A, Mark J, Zender C, Gillenwater AM, Bell D, Kurtzweil N, Mathews M, Allen CL, Mierzwa ML, Casper K, Jandarov R, Medvedovic M, Lee JJ, Harun N, Takiar V, Gillison M. Phase II Clinical Trial of Neoadjuvant and Adjuvant Pembrolizumab in Resectable Local-Regionally Advanced Head and Neck Squamous Cell Carcinoma. Clin Cancer Res. 2022 Apr 1;28(7):1345-1352. doi: 10.1158/1078-0432.CCR-21-3351. PMID 35338369
- [Background] Uppaluri R, Campbell KM, Egloff AM, Zolkind P, Skidmore ZL, Nussenbaum B, Paniello RC, Rich JT, Jackson R, Pipkorn P, Michel LS, Ley J, Oppelt P, Dunn GP, Barnell EK, Spies NC, Lin T, Li T, Mulder DT, Hanna Y, Cirlan I, Pugh TJ, Mudianto T, Riley R, Zhou L, Jo VY, Stachler MD, Hanna GJ, Kass J, Haddad R, Schoenfeld JD, Gjini E, Lako A, Thorstad W, Gay HA, Daly M, Rodig SJ, Hagemann IS, Kallogjeri D, Piccirillo JF, Chernock RD, Griffith M, Griffith OL, Adkins DR. Neoadjuvant and Adjuvant Pembrolizumab in Resectable Locally Advanced, Human Papillomavirus-Unrelated Head and Neck Cancer: A Multicenter, Phase II Trial. Clin Cancer Res. 2020 Oct 1;26(19):5140-5152. doi: 10.1158/1078-0432.CCR-20-1695. Epub 2020 Jul 14. PMID 32665297